CLINICAL TRIAL: NCT05633173
Title: Comparison of the Effects of Erector Spinae Plane Block and Caudal Block on Postoperative Analgesia and Stress Response in Pediatric Patients Undergoing Inguinal Hernia Surgery, Prospective Randomized Trial
Brief Title: Effects of Erector Spinae Plane and Caudal Block on Postoperative Stress Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Özge Uyanıkoğlu, Medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7931
Record Dates: First submitted 2022-11-17; First posted 2022-12-01 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Post Operative Pain; Stress Response; Erector Spinae Plane Block; Caudal Block
Keywords: Pediatric regional anesthesia; Erector spina plane block; Caudal block; Surgical stress hormone
MeSH Terms: conditions — Pain, Postoperative; Fractures, Stress

STUDY DESIGN:
Intervention Model Description: The patients to be included in the study were randomized into two groups, Group E and C, using the closed envelope method in the preoperative period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Experimental): Ultrasound-guided erector spina plan block was performed for patients in group E for postoperative analgesia. The patients were placed in the lateral decubitus position and the linear ultrasound probe was placed longitudinally into the sterilized area 1-2 cm lateral to the spinous process of the L1 vertebra. After visualizing the erector spina muscle and the transverse process, the transverse process was reached by pushing forward the 22 gauge, 50 mm needle in the direction from cranial to caudal. Hydrodissection was performed with 1 ml of saline for confirmation. 0.5 mL kg-1 dose of 0.25% bupivacaine was injected under the erector spina muscle at the level of the 1st lumbar vertebra by aspiration every 2 mL.
  Interventions: Procedure: Ultrasound-guided erector spinae plan block
- Group C (Active Comparator): The patients in group C underwent ultrasound guided caudal block for postoperative analgesia. By placing the patients in the lateral decubitus position, the linear ultrasound probe was placed longitudinally on the sterilized area on the midline of the sacrum, and access was provided with a 2.5 cm 22 gauge needle on the dorsal skin of the sacral hiatus at a 90° position. The sacrococcygeal ligament was crossed, the needle was oriented approximately 25° and advanced approximately 2 to 3 mm to reach the sacral canal. When it was understood that the sacral hiatus had been entered, 0.5 mL kg-1 0.25% bupivacaine was injected by aspirating every 2 mL after the location was confirmed with the negative aspiration method.
  Interventions: Procedure: Ultrasound-guided caudal block

INTERVENTIONS:
Procedure: Ultrasound-guided erector spinae plan block — Ultrasound-guided erector spina plan block was performed for patients in group E for postoperative analgesia. The patients were placed in the lateral decubitus position and the linear ultrasound probe was placed longitudinally into the sterilized area 1-2 cm lateral to the spinous process of the L1 vertebra. After visualizing the erector spina muscle and the transverse process, the transverse process was reached by pushing forward the 22 gauge, 50 mm needle in the direction from cranial to caudal. Hydrodissection was performed with 1 ml of saline for confirmation. 0.5 mL kg-1 dose of 0.25% bupivacaine was injected under the erector spina muscle at the level of the 1st lumbar vertebra by aspiration every 2 mL.
  Arms: Group E
Procedure: Ultrasound-guided caudal block — The patients in group C underwent ultrasound guided caudal block for postoperative analgesia. By placing the patients in the lateral decubitus position, the linear ultrasound probe was placed longitudinally on the sterilized area on the midline of the sacrum, and access was provided with a 2.5 cm 22 gauge needle on the dorsal skin of the sacral hiatus at a 90° position. The sacrococcygeal ligament was crossed, the needle was oriented approximately 25° and advanced approximately 2 to 3 mm to reach the sacral canal. When it was understood that the sacral hiatus had been entered, 0.5 mL kg-1 0.25% bupivacaine was injected by aspirating every 2 mL after the location was confirmed with the negative aspiration method.
  Arms: Group C

SUMMARY:
Inguinal hernia surgery is the most common practice of pediatric surgeons in their clinical practice. As these operations are usually day case procedures, maintaining adequate analgesia is an important component of perioperative care and ERAS protocols. Caudal block, which is one of the analgesic methods used for postoperative pain, is the most frequently used in inguinal hernia surgery and its effectiveness has been proven. Erector spina plane block, which is easy to apply and has a low risk of side effects, is another tool used in the treatment of postoperative pain after inguinal hernia surgery. These are the procedures that are routinely applied in our center with the aim of intraoperative and postoperative effective analgesia.

DETAILED DESCRIPTION:
Surgery is a common medical procedure that exposes children to pain. More than 85% of children experience clinically significant pain after surgery and 63% after discharge. Postoperative pain management in pediatric ages also plays a role in future pain perception and chronic pain development. It has been reported that acute postoperative pain progresses to chronic pain in 20% of children undergoing major surgery. It is also known that children with inadequate pain management experience a decline in immune and neuroendocrine functions later in life.

Inguinal hernia surgery is one of the most frequently performed elective surgeries in pediatric surgery practice and often performed in early childhood. The presence of postoperative pain delays the return to normal activity and prolongs the time to discharge. Ideal pain management should provide complete pain relief without interfering with the child's daily life, and the techniques and drugs used in the treatment should cause as few side effects as possible. Opioid and non-opioid analgesics have side effects such as itching, vomiting, delay in gastrointestinal function, urinary retention, respiratory depression, liver failure, antithrombotic effect, delayed wound healing, renal and gastrointestinal toxicity that limit their use in children.

In recent years, multimodal analgesia in which non-opioid analgesics are combined with small doses of opioids or regional blocks is increasingly preferred. Caudal block, one of the regional blocks, has been widely used in pediatric surgery for many years due to its proven effectiveness in postoperative analgesia. In addition, with the widespread use of ultrasound, many body blocks have become used with high success rates in both upper and lower abdominal surgeries in postoperative pain management. Erector spina plane block (ESPB), defined by Forrero et al. in 2016, is an interfacial plane block that is a simpler and safer alternative to thoracic epidural or paravertebral block. Its use for analgesia is common in adults in various surgeries, and its use in pediatric surgeries is also becoming widespread. In a review published in 2019, it was reported that only 23 of 242 ESPB cases were children. Clinical studies of ESPB applied in pediatric patients are not sufficient in the literature.

Tissue damage caused by surgery or trauma brings hormonal, metabolic and hemodynamic changes. It is known that post-surgical stress response causes major changes in the cardiovascular and respiratory systems. Controlling postoperative pain is associated with decreased stress hormone response. The scales used in the evaluation of postoperative pain in pediatric patients are insufficient due to the inability of the patients to express themselves and their high anxiety coefficients. For this reason, it has been suggested that stress hormone levels may be an objective method for determining the analgesic efficacy of the anesthetic technique. Early mobilization and postoperative pain management gain importance in inguinal hernia surgery, since they are outpatient surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) class I-II patients
* Patients aged 1 - 6 years
* Patients who will undergo unilateral inguinal hernia surgery

Exclusion Criteria:

* ASA III - IV patients
* Emergency surgery patients
* Children of parents who did not give consent
* Patients with chronic pain
* Local anesthetic allergy
* Infection in the block area
* Coagulopathy
* Increased intracranial pressure
* Neurological deficit
* Severe organ failure
* Mental retardation
* Anatomical deformities

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Stress Response | 3 hours
  serum concentration of Cortisol, serum concentration of Prolactin

SECONDARY OUTCOMES:
FLACC scores | 24 hours
  Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Pain Scale. FLACC is abehavioral pain assessment scale used for nonverbal or preverbal patients who areunable to self-report their level of pain. Pain is assessed through observation of 5categories including face, legs, activity, cry, and consolability. The increase in thepain felt by the patient also increases the fl acc score. Each category is scored onthe 0-2 scale which results in a total score of 0-10.
Analgesic Consumption | 24 hours
  The total amount of analgesic in the first 24 hours
Analgesia Time | 24 hours
  The time of first analgesic need
Complications | 24 hours
  Hypotension, bradycardia, vomiting, itching

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Surhan ÇINAR, Study Chair — Sisli Hamidiye Etfal Research and Training Hospital
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No